CLINICAL TRIAL: NCT01830751
Title: Influencing Diurnal Variation in Disc Hydration as a Treatment for Non-specific Low Back Pain
Brief Title: Limiting Trunk Flexion as a Self-treatment for Low Back Pain
Acronym: RST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liberty Mutual Research Institute for Safety (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LMRIS 12-02
Record Dates: First submitted 2013-03-29; First posted 2013-04-12 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Low Back Pain
Keywords: self treatment technique; chronic; non specific; LBP; control trunk flexion; diurnal
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Limit trunk flexion upon rising (Experimental): Immediately upon rising particpants perform the Restrained Sitting Treatment intervention for one hour.
  Interventions: Other: Restrained Sitting Treatment
- Limit trunk flexion before going to bed (Sham Comparator): Immediately prior to going to bed, particpants perform the Restrained Sitting Treatment intervention for one hour.
  Interventions: Other: Restrained Sitting Treatment

INTERVENTIONS:
Other: Restrained Sitting Treatment — Training in avoidance of trunk flexion, with the use of a tall backrest with lumbar support to which the participant straps themselves. Participants are taught to strap into the backrest while while seated in a chair, and with hips and knees bent at right angles, for one hour at the appointed time of day.

SUMMARY:
The purpose of the proposed study is to test the effect of an intervention technique that reduces trunk flexion upon rising, on the outcome measures of self-reported back pain and functional impairment in individuals with chronic or recurrent non-specific low back pain (LBP). The intervention is a self-administered and requires no medical intervention or drugs. The technique referred to as the restrained sitting treatment (RST), involves training in minimizing forward bending of the trunk immediately upon rising. The technique builds upon a previous randomized controlled study conducted and published by members of the research team. The underlying premise of RST exploits the natural diurnal pattern as the intervertebral discs (people are tallest when they first wake up). The discs are fully hydrated upon rising, disc internal hydrostatic pressures and external forces acting on surrounding soft tissues are greatest at this time, and these pressures and forces can increase significantly with trunk flexion. The RST technique utilizes a back support used in sitting during the first hour upon rising to minimize trunk flexion during this critical period as the intervertebral discs begins the diurnal cycle of fluid loss. The study will test the null hypothesis that there are no significant difference in outcome (LBP, work or social function/disability) between groups performing RST, the experimental group performing RST upon rising, the control group performing prior to going to bed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic or recurrent low back pain
* Six month or longer history of non-specific LBP
* Minimum 90 days in pain in the last six months
* Average pain score of past month ≥3 on a 0-10 numerical rating scale

Exclusion Criteria:

* Red flags (tumor, metabolic diseases, Rheumatoid arthritis, osteoporosis, prolonged steroid use, pregnancy, back surgery)
* Evidence of nerve root compression (pain reproduction with SLR>45º, weakness of major lower extremity muscle group, decreased deep tendon reflexes at knee or ankle, decreased sensation to pinprick)
* Acute trauma to low back

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Pain Score (numerical rating scale 0-10) | Baseline and 3 months (end of intervention phase)
  Change in mean number of days reporting disability from beginning to end of intervention phase

SECONDARY OUTCOMES:
Functional limitation in work | Baseline and 3 months (end of intervention phase)
  Change in mean number of days reporting disability from beginning to end of intervention phase
Medication taken for back pain | Baseline and 3 months (end of intervention phase)
  Change in mean number of days reporting medication use from beginning to end of intervention phase

CONTACTS AND LOCATIONS:
Overall Officials: Raymond W McGorry, MS, PT, Principal Investigator — Liberty Mutual Research Institute for Safety
Locations (1):
- Liberty Mutual Research Institute for Safety, Hopkinton, Massachusetts, United States